CLINICAL TRIAL: NCT05182502
Title: A Prospective, Single-center, Single-arm Clinical Study Evaluating the Safety and Effectiveness of the Tixel Fractional System in the Treatment of Photodamage at Low Settings
Brief Title: Evaluating the Safety and Effectiveness of the Tixel Fractional System in the Treatment of Photodamage at Low Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eric Bernstein, MD (Other)
Collaborators: Novoxel Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Eric Bernstein, MD, Principal Investigator, Main Line Center for Laser Surgery
Organization: Main Line Center for Laser Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tixel2021
Record Dates: First submitted 2021-12-16; First posted 2022-01-10 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Wrinkle
Keywords: wrinkle; photo damage

STUDY DESIGN:
Intervention Model Description: Treatment of subjects with a device for facial rejuvenation and blinded comparison of pre- and post-treatment photos.
Masking Description: Photos will be evaluated in randomized blinded pairs pre- and post-treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tixel treatment arm (Experimental): subjects will receive 3 monthly treatments with the Tixel device
  Interventions: Device: Tixel

INTERVENTIONS:
Device: Tixel — Subjects will receive 3 monthly treatments with the Tixel device to treat the signs of photodamage

SUMMARY:
To demonstrate the safety and performance of the Tixel fractional system for treatment of photodamage using low-energy settings.

DETAILED DESCRIPTION:
A Prospective, single-center, single-arm clinical study of subjects who are seeking a procedure to reduce the appearance of photodamage, and meet study eligibility criteria, and have provided informed consent will be enrolled in the study. One investigational center will participate in the recruitment. Each study subject will receive 3 treatments with Tixel at 4-6 week intervals. Final follow-up will occur 3 months following the last treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 25-70 years old with clinically evident photodamage.
2. Willingness and ability to comply with all required study activities including returning for follow-up visits and protocol requirements.
3. The subject is able to provide written informed consent and perform the study's activities according to HIPAA guidelines.
4. Fitzpatrick wrinkle score of 3-7 in the per the treating investigator and clinically noticeable wrinkles in the treating area.
5. Skin Type I - V as per Fitzpatrick Skin Scale.

Exclusion Criteria:

1. Past treatment with Tixel device.
2. The subject may not undergo treatment by the Tixel device according to the device's contra-indications for use, as defined in the User Manual and in the Instructions for Use and by any other labeling of the device.
3. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
4. Female subjects who are pregnant or planning to become pregnant.
5. Subjects with significant exposure to critical amounts of ultraviolet light (Suntan).
6. Subjects who have had the following treatments:

   1. a cosmetic procedure to improve rhytides (i.e. Carbon Dioxide/Erbium/similar laser/fractional resurfacing, radiofrequency treatment) within 3 months
   2. prior facial treatments with laser, surgical, chemical or light-based facial treatments within the previous 3 months, including botulinum toxin injections or microdermabrasion.
   3. Injectable filler in cheeks (mid face) temples and in the upper face area to be treated within 3 months of investigation.
7. Any subject who has visible scars or other visible changes over the treated areas that may affect evaluation of response and/or quality of photography.
8. Subjects with any type of active cut, wound, inflammation, premalignant or malignant lesion or active bacterial, viral, fungal, or herpetic infection on the skin on the designated treatment sites or in close proximity to it.
9. Existing or history of the following (when discussing skin conditions, refers only to the face):

   1. skin malignancy, or any diagnosis of suspected malignancy
   2. Collagen vascular or bleeding disorder
   3. Immunosuppression or autoimmune disease
   4. Active acne vulgaris, herpes simplex virus or any existing skin condition/disease that in the investigator's opinion would interfere with the evaluation of the safety of the study treatment and evaluation.
   5. Any skin pathology which can induce bullous lesions, urticaria, or demonstrate a Koebner phenomenon (psoriasis, lichen planus, etc.).
   6. Any disease that inhibits pain sensation
   7. History of keloid formation, or hypertrophic scarring
   8. Conditions affecting healing rate (diabetes mellitus I or II)
   9. neuromuscular disorders
10. Subjects who have used, within 30 days, any medication that can cause dermal hypersensitivity or affect skin characteristics over the treated area (i.e. topically applied retinoids, hydroquinone, chemical peel of any strength: glycolic acid, lactic acid, salicylic acid)
11. Subjects who have used, systemic treatment which may induce dyspigmentation, such as amiodarone, clofazimine, or chloroquine.
12. Subjects currently taking or have taken an oral retinoid in the past six months; Subjects currently taking long-term oral corticosteroid treatment.
13. Concurrent therapy that, in the principal investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study treatment.
14. Subjects who anticipate the need for major surgery or overnight hospitalization during the study that can affect the study schedule or treatment evaluation.
15. Enrollment in any active study involving the use of investigational devices or drugs.
16. Any other cause per the principal investigator's discretion.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Blinded photo evaluation | 3 months post-treatment
  blinded observer rating of photos for photo damage using the Fitzpatrick Wrinkle Classification Scale: Class Description Score Description I Fine wrinkles 1-3 Mild: Fine texture changes with subtly accentuated skin lines.
  II Fine to moderate depth wrinkles, Moderate number of lines 4-6 Moderate: Distinct papular elastosis (individual papules with yellow translucency under direct lighting) and dyschromia III Fine to deep wrinkles, numerous lines, with or without redundant skin folds 7-9 Severe: Multipapular and confluent elastosis (thickened, yellow, and pallid) approaching or consistent with cutis rhomboidalis.

CONTACTS AND LOCATIONS:
Overall Officials: Eric F. Bernstein, MD, Principal Investigator — Main Line Center for Laser Surgery
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No